CLINICAL TRIAL: NCT00000339
Title: Infusion Laboratory: Protocol 3 (Risperidone)
Brief Title: Infusion Laboratory: Protocol 3 (Risperidone) - 4
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: NIDA-3-0010-4; Y01-3-0010-4
Record Dates: First submitted 1999-09-20; First posted 1999-09-21 (Estimated); Last update posted 2017-01-11 (Estimated); Status verified 1996-06

CONDITIONS: Cocaine-Related Disorders
Keywords: cocaine dependence
MeSH Terms: conditions — Cocaine-Related Disorders | interventions — Risperidone

INTERVENTIONS:
Drug: Risperidone

SUMMARY:
The purpose of this study is to evaluate clinical safety issues pertaining to risperidone, to cocaine and to its interaction, and to determine how pretreatment with risperidone modifies the subjective as well as physiological effects of cocaine.

ELIGIBILITY:
Inclusion Criteria:

M/F ages 21-50. Meet DSM-IV criteria for cocaine dependence. Agree to conditions of the study and sign informed consent.

Exclusion Criteria:

Psychiatric disorder that requires medication therapy. History of seizures. Pregnant and/or nuring women. Dependence on ETOH or benzodiazepines or other sedative/hypnotics. Acute hepatitis. Other medical condtions that deem participation to be unsafe.

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 13
Dates: Start 1996-06

PRIMARY OUTCOMES:
Evidence of change in neurotoxicity based on chore
Degree of drug craving
History, incidence and amount of drug use
Type and severity of stimulant withdrawal symptoms
Characterization of study population
Population incidence of symptoms of depression, po
Frequency and intensity of drug use and sexual beh
Evidence of change in subjective responses to coca
Clinical physiological response to cocaine challen
Degree to which study medication influences change

CONTACTS AND LOCATIONS:
Overall Officials: Walter Ling, M.D., Principal Investigator — Friends Research Institute, Inc.
Locations (1):
- Friends Research Institute, Los Angeles, California, United States